CLINICAL TRIAL: NCT05888168
Title: A Comprehensive Observational Study on the Determinants of Postoperative Atrial Fibrillation in Patients Undergoing Coronary Artery Bypass Grafting
Brief Title: Predictors of Postoperative Atrial Fibrillation After CABG
Acronym: CODA-AF
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Kun Hua (Other)
Responsible Party: Sponsor-Investigator, Kun Hua, Deputy Chief Surgeon, Beijing Anzhen Hospital
Organization: Beijing Anzhen Hospital (Other)
Other Study IDs: 2023065X
Record Dates: First submitted 2023-05-21; First posted 2023-06-05 (Actual); Last update posted 2023-06-05 (Actual); Status verified 2023-06

CONDITIONS: Coronary Artery Disease; Atrial Fibrillation New Onset
Keywords: coronary artery bypass grafting; postoperative atrial fibrillation
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- POAF: This group will consist of patients who have developed postoperative atrillary fibrillation (POAF) after undergoing coronary artery bypass grafting (CABG).
  Interventions: Procedure: CABG
- Non-POAF: This group will consist of patients who have not developed postoperative atrillary fibrillation (POAF) after undergoing coronary artery bypass grafting (CABG).
  Interventions: Procedure: CABG

INTERVENTIONS:
Procedure: CABG — All participants in the study will undergo the standard procedure of CABG. Continuous electrocardiogram monitoring and electrocardiography were used to identify the cardiac rhythm.

SUMMARY:
This observational study aims to identify the determinants or predictors of postoperative atrial fibrillation (POAF) in patients who have undergone coronary artery bypass grafting (CABG). The study will compare two cohorts: patients who developed POAF and those who did not (non-POAF), with the aim of improving postoperative care, reducing complications, and refining patient risk stratification.

DETAILED DESCRIPTION:
Demographics (age, sex, ethnicity), lifestyle factors (smoking, alcohol, physical activity), and medical history (diabetes, hypertension, prior heart diseases) will be recorded. Surgical procedure details (number of grafts, use of intraoperative devices), anesthesia, and medications administered. Levels of inflammatory markers, cardiac-specific markers, and other relevant biomarkers at baseline and postoperatively. Other complications besides POAF, hospital length of stay, ICU admission, readmission rate, and mortality will also be monitored.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 18 years or older.
* Patients who underwent CABG.

Exclusion Criteria:

* Patients with a history of preoperative atrial fibrillation or other significant arrhythmias.
* Patients who underwent other concurrent cardiac procedures (e.g., valve surgery) in addition to CABG.
* Patients who cannot provide informed consent or lack adequate follow-up information.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The participants in this study are adult patients (18 years and older) who have undergone Coronary Artery Bypass Grafting (CABG). These individuals come from diverse demographic backgrounds and have a history of severe coronary heart disease, the condition that necessitated the CABG surgery.
Sampling Method: Non-Probability Sample
Enrollment: 15000 (Estimated)
Dates: Start 2018-01-01 (Actual); Primary Completion 2023-12-15 (Estimated); Study Completion 2024-05-01 (Estimated)

PRIMARY OUTCOMES:
Incidence of POAF | During hospital stay, up to 30 days
  This will be determined based on electrocardiograms (ECG) and/or relevant medical records, within 30 days post-CABG.

SECONDARY OUTCOMES:
Hospital length of stay | During hospital stay, up to 30 days
ICU admission time | During hospital stay, up to 30 days
Number of participants with Stroke | During hospital stay, up to 30 days
Mortality | During hospital stay, up to 30 days

CONTACTS AND LOCATIONS:
Overall Officials: Kun Hua, MD, Study Chair — Beijing Anzhen Hospital
Locations (1):
- Beijing Anzhen Hospital, Beijing, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Zhou X, Pan Y, Hua K, Yang X. Impact of Sodium-Glucose Cotransporter 2 Inhibitors on Acute Kidney Injury Post Off-Pump Coronary Artery Bypass Grafting: A Retrospective Cohort Study and Meta-Analysis. Rev Cardiovasc Med. 2026 Jan 21;27(1):39400. doi: 10.31083/RCM39400. eCollection 2026 Jan. PMID 41659092